CLINICAL TRIAL: NCT00755937
Title: Remicade® Treatment Registry Across Canada in Crohn's Disease
Brief Title: Remicade® Crohn's Disease Registry Across Canada (Study P02793)
Acronym: RemiTRAC®
Status: Terminated | Type: Observational
Why Stopped: Satisfied a post-marketing commitment to Canadian Health Authorities.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P02793
Record Dates: First submitted 2008-08-26; First posted 2008-09-19 (Estimated); Results first posted 2009-06-11 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects receiving Remicade: Crohn's disease subjects receiving Remicade® per Product Monograph.
  Interventions: Other: Data collection post infusion

INTERVENTIONS:
Other: Data collection post infusion

SUMMARY:
This registry is a multi-center, prospective, observational program that will gather and analyze data on subjects with Crohn's disease being treated with Remicade® as per approved product monograph in Canada. In contrast to a controlled clinical trial, there is no imposed experimental intervention and treatment with Remicade® is determined solely by the subject's physicians. Thus, the data captured and reported in this registry will reflect a "real world" approach to the treatment of Crohn's disease with Remicade®.

DETAILED DESCRIPTION:
Subjects will be selected for this registry using a non-probability sampling method.

ELIGIBILITY:
Inclusion Criteria:

* Patient was given the Patient Information Brochure; AND,
* Patient has never been treated with Remicade® (patient is naïve to Remicade® at the time of registration); AND,
* Patient is a good candidate to receive Remicade® as per the product monograph; AND,
* Patient has agreed to complete the Patient Diary for one week prior to each visit in the registry; AND,
* Patient has signed the approved consent form.

Exclusion Criteria:

* Per product monograph

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primarily from community centers and some academic centers.
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2002-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational trial/registry. Recruitment began in 2002. Subjects were drawn from community centers and some academic centers.
Pre-assignment Details: Not applicable for an observational trial. Subjects were not assigned to treatment, but received infliximab only if their physician had decided to treat with infliximab.
Groups:
- Subjects Receiving Remicade: Crohn's disease subjects who were to receive Remicade® per Product Monograph.
Period: Recruitment
Arm/Group | Subjects Receiving Remicade
Started | 556 (Subjects registered in the program)
Completed | 392 (Subjects who had a baseline visit and at least 1 additional follow-up visit (analyzed population))
Not Completed | 164
Not completed — Unknown if infliximab received | 164
Period: Observational Follow-up
Arm/Group | Subjects Receiving Remicade
Started | 392
Completed | 244 (Subjects followed until end of study/subjects for whom end of participation data were collected)
Not Completed | 148
Not completed — Lost to Follow-up | 148

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Receiving Remicade
Number analyzed (Participants) | 556
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314
  Male | 242
Region of Enrollment [Number; unit: participants]
  Canada | 556

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at 12 Months (Decrease in Crohn's Disease Activity Index [CDAI]>= 70 Points AND >= 25% From Baseline).
Description: CDAI is calculated based on 8 factors: # of liquid stools, abdominal pain, patient well-being, Crohn's complications, need for anti-diarrheal medications, abdominal mass, hematocrit, and weight. CDAI can range from 0 to 600. Remission is < 150, and moderate to severe disease ranges from 220 to 450.
Time Frame: 12 months after baseline
Population: Patients at 12 months: Patients with at least 12 months of follow-up. Imputation for missing values used either the last observation carried forward or last observation carried backward, whichever had the highest CDAI.
Measure: Number; unit: Participants
Arm/Group | Subjects Receiving Remicade
Number analyzed (Participants) | 179
Participants | 118
Statistical Analysis 1: Comparison: Subjects Receiving Remicade; Test type: Superiority or Other; There were no comparisons between groups as this was a single-arm observational study; Percentage (no inferential test) = 66.3

2. Primary Outcome: Clinical Response at 24 Months (Decrease in CDAI >= 70 Points AND >= 25% From Baseline).
Description: as for outcome 1
Time Frame: 24 months after baseline
Population: Patients at 24 months: Patients with at least 24 months of follow-up. Imputation for missing values used either the last observation carried forward or last observation carried backward, whichever had the highest CDAI.
Measure: Number; unit: Participants
Arm/Group | Subjects Receiving Remicade
Number analyzed (Participants) | 91
Participants | 66
Statistical Analysis 1: Comparison: Subjects Receiving Remicade; Test type: Superiority or Other; There were no comparisons between groups as this was a single-arm observational study; percentage (no inferential test) = 72.5

3. Primary Outcome: Clinical Response at 36 Months (Decrease in CDAI >= 70 Points AND >= 25% From Baseline).
Description: as for outcome 1
Time Frame: 36 months after baseline
Population: Patients at 36 months: Patients with at least 36 months of follow-up. Imputation for missing values used either the last observation carried forward or last observation carried backward, whichever had the highest CDAI.
Measure: Number; unit: Participants
Arm/Group | Subjects Receiving Remicade
Number analyzed (Participants) | 43
Participants | 31
Statistical Analysis 1: Comparison: Subjects Receiving Remicade; Test type: Superiority or Other; There were no comparisons between groups as this was a single-arm observational study; Percentage (no inferential test) = 72.1

4. Primary Outcome: Clinical Remission at 12 Months (CDAI <= 150 Points).
Description: as for outcome 1
Time Frame: 12 months after baseline
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Subjects Receiving Remicade
Number analyzed (Participants) | 179
Participants | 108
Statistical Analysis 1: Comparison: Subjects Receiving Remicade; Test type: Superiority or Other; There were no comparisons between groups as this was a single-arm observational study; Percentage (no inferential test) = 60.3

5. Primary Outcome: Clinical Remission at 24 Months (CDAI <= 150 Points).
Description: as for outcome 1
Time Frame: 24 months after baseline
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Subjects Receiving Remicade
Number analyzed (Participants) | 91
Participants | 59
Statistical Analysis 1: Comparison: Subjects Receiving Remicade; Test type: Superiority or Other; There were no comparisons between groups as this was a single-arm observational study; Percentage (no inferential test) = 64.8

6. Primary Outcome: Clinical Remission at 36 Months (CDAI <= 150 Points).
Description: as for outcome 1
Time Frame: 36 months after baseline
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Subjects Receiving Remicade
Number analyzed (Participants) | 43
Participants | 31
Statistical Analysis 1: Comparison: Subjects Receiving Remicade; Test type: Superiority or Other; There were no comparisons between groups as this was a single-arm observational study; Percentage (no inferential test) = 72.1

7. Secondary Outcome: Number of Serious Adverse Events
Time Frame: Throughout study (up to 36 months)
Population: Safety data were collected for all patients registered. Total number of subjects: 556. Non serious adverse events: 198. Serious Adverse Events: 105.
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Subjects Receiving Remicade
Number analyzed (Participants) | 556
Number of Serious Adverse Events | 105

ADVERSE EVENTS:
Description: Subjects who had a baseline visit and at least 1 additional follow-up visit (analyzed population) were included in this analyses.
Arm/Group | Subjects Receiving Remicade
Serious Adverse Events (participants affected / at risk) | 39/392
Other Adverse Events (participants affected / at risk) | 0/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Receiving Remicade (N=392)
PALPITATIONS (Cardiac disorders) | 1 (1)
EYE OEDEMA (Eye disorders) | 1 (1)
RETINAL DISORDER (Eye disorders) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3)
APPENDICITIS PERFORATED (Gastrointestinal disorders) | 1 (1)
CROHN'S DISEASE (Gastrointestinal disorders) | 10 (11)
DIARRHOEA (Gastrointestinal disorders) | 1 (2)
FAECALOMA (Gastrointestinal disorders) | 1 (1)
ILEAL STENOSIS (Gastrointestinal disorders) | 1 (1)
INTESTINAL STENOSIS (Gastrointestinal disorders) | 1 (1)
PERITONITIS (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 (3)
VOMITING (Gastrointestinal disorders) | 1 (1)
CHEST PAIN (General disorders) | 1 (1)
DEATH (General disorders) | 1 (1)
DRUG INEFFECTIVE (General disorders) | 2 (2)
FATIGUE (General disorders) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 2 (2)
PYREXIA (General disorders) | 1 (1)
THERAPEUTIC RESPONSE DECREASED (General disorders) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 2 (2)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1)
BRAIN ABSCESS (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 1 (1)
MENINGITIS VIRAL (Infections and infestations) | 1 (1)
PERIANAL ABSCESS (Infections and infestations) | 2 (2)
RECTAL ABSCESS (Infections and infestations) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1)
TOOTH ABSCESS (Infections and infestations) | 1 (1)
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 1 (1)
DRUG EXPOSURE DURING PREGNANCY (Injury, poisoning and procedural complications) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
MENTAL DISORDER (Psychiatric disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BLISTER (Skin and subcutaneous tissue disorders) | 1 (1)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1)
PROCTOCOLECTOMY (Surgical and medical procedures) | 1 (1)
SURGERY (Surgical and medical procedures) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an observational study. There were no imposed interventions from the Sponsor including imposing specific duration of treatment or data collection beyond the standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No